CLINICAL TRIAL: NCT05690841
Title: FocaL Mass Drug Administration for Vivax Malaria Elimination (FLAME): a Pragmatic Cluster Randomized Controlled Trial in Peru
Brief Title: FocaL Mass Drug Administration for Vivax Malaria Elimination
Acronym: FLAME
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Universidad Peruana Cayetano Heredia- subcontractor to UCSF as local Sponsor (Unknown); PATH (Other); Stanford University (Other); Oxford University Clinical Research Unit Indonesia (Other); Menzies School of Health Research (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-36417; 1U01AI157962 (NIH); 23-0008 (Other: UCSF IRB)
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Plasmodium Vivax Malaria; Malaria
Keywords: Antimalarial drugs; Primaquine; Chloroquine; Tafenoquine; Parasitic disease
MeSH Terms: conditions — Malaria, Vivax; Malaria; Parasitic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control: Standard Interventions (No Intervention): Standard interventions for the control cluster will include providing participants with long-lasting insecticide-treated bednets, management of known and possible mosquito breeding sites, passive case detection through detection and diagnosis of symptomatic cases of malaria in health facilities and through community health workers (conducted in villagers with fever), microscopy testing in households of recent index cases to detect asymptomatic malaria cases, and treatment of active cases of malaria (artesunate-mefloquine (AS-MQ) for Plasmodium falciparum and Chloroquine (CQ) (10 mg/kg on days 1 and 2, followed by 5 mg/kg on day 3) + PQ (0.5mg/kg x 7 days).
- Focal Mass Drug Administration (fMDA) (Experimental): Standard interventions in addition to focal mass drug administration. Focal mass drug administration will include using primaquine, chloroquine, and tafenoquine, for high-risk individuals residing in households that are within 200 meters of a Plasmodium vivax (Pv) index case households from the prior 2 years (including individuals in the index case household). Pv index cases include symptomatic cases detected at health facilities or in fever screenings, and asymptomatic cases identified during routine active case detection by health facilities. Households will then be notified regarding their potential to receive two rounds fMDA that cycle. Eligibility to receive medications as part of fMDA will be assessed prior to each administration and include glucose 6 phosphate dehydrogenase (G6PD) testing and counseling if not previously conducted or result is not available on the participant's identification card.
  Interventions: Drug: Focal Mass Drug Administration (fMDA)

INTERVENTIONS:
Drug: Focal Mass Drug Administration (fMDA) — Administration of focal mass drug administration for high-risk individuals residing in households that are within 200 meters of a Plasmodium vivax index case households from the prior 2 years (including individuals in the index case household). Intervention to be administered two times, two months apart each cycle, for 3 cycles spaced apart by regular intervals.
  Each year will include 2 rounds of fMDA.
  Round 1) Chloroquine (CQ)+ Tafenoquine (TQ) for >= 16y (CQ: Day1 600 mg, Day 2 600 mg, Day 3 300 mg CQ, TQ 300 mg on Day 1); CQ+ Primaquine (PQ) for <16y (CQ: age-based dosing, PQ age-based dosing); CQ+PQ for G6PD intermediate individuals >=6mo and <16y ((CQ: Day1 600 mg, Day 2 600 mg, Day 3 300 mg, PQ age-based dosing).
  Round 2) single dose CQ+TQ for >= 16y (CQ: Day1 600 mg, TQ 300 mg on Day 1); single dose CQ+PQ for <16y (CQ: age-based dosing, PQ age-based dosing); single dose CQ+PQ for G6PD intermediate individuals >=6mo and <16y ((CQ: Day1 600 mg, PQ age-based dosing).
  Arms: Focal Mass Drug Administration (fMDA)

SUMMARY:
FLAME is an open-label cluster-randomized controlled trial that aims to determine the effectiveness of focal mass drug administration (fMDA) to reduce the incidence of Plasmodium vivax malaria in the Loreto Department in Peru. Standard interventions, including symptomatic and asymptomatic screening for malaria infections, provision of insecticide-treated bednets, and environmental transmission monitoring, will be compared to clusters of villages randomized to receive anti-malarial drugs.

DETAILED DESCRIPTION:
This trial is an open-label cluster-randomized controlled trial in Loreto Region, Peru, a low transmission setting (i.e. anual incidence <250/1000), where the unit of randomization is a village, or cluster. There will be two study arms: Control and fMDA. Villages will receive fMDA or control based on a restricted randomization that includes baseline factors such as incidence, distance to a health post, and population.

The interventions for both control and fMDA clusters will include standard interventions (high coverage of vector control, passive and active symptomatic case management, and RACD of asymptomatic cases). The intervention will take place in 2 rounds for three cycles, each cycle separated by regular intervals. fMDA will target high-risk villagers (individuals residing in households that are within 200 meters of a Pv index case households from the prior 2 years). High-risk status will be determined in each survey before the administration of Round "a" of fMDA. Pv index cases refers to confirmed Pv cases reported by the health system.

In each cycle of fMDA, the 1st round will include 3 days of chloroquine (CQ) for treatment of Pv asexual blood stages, with TQ for Pv liver stages. With a prolonged half-life up to 15 days and post-treatment effect observed up to 77 days. TQ will also have a prophylactic and likely gametocytocidal effect for Pv and Pf. For continued anti-relapse, prophylactic, and transmission-blocking effects, a follow-up round will include TQ with single-dose CQ (sdCQ). If TQ, but not PQ, is contraindicated, a standard 7-day PQ course will be used. CQ, including in a single dose, will potentiate the anti-relapse effect of PQ, and likely TQ. Preliminary data from the study area shows that 32% of the study population is <16 years old and will receive PQ. However, the investigators do not anticipate this to influence the impact of the fMDA due to our use of directly observed therapy (DOT). If pediatric TQ is approved for use in Peru during the study, an addendum to the protocol will be presented for approval by the IRB and INS and incorporated into the study.

An endline survey will be carried out at the end of the 3-year trial intervention period. An interim survey will also be conducted in a subset of the population both arms. In each of these surveys, a dried blood spot will be collected from all participants. Anyone with fever in the prior 48 hours and a positive blood smear from a local health post will receive treatment per national policy. Anyone with fever in the prior 48 hours without a positive blood smear will be encouraged to go to a health post. To maximize public health relevance, the trial will be pragmatic and implemented through the existing health system.

The primary research objectives are:

1. To determine the effectiveness of three rounds of fMDA to reduce Pv transmission in the Loreto Department, Peru compared to standard interventions.
2. To evaluate the safety and tolerability of fMDA by measuring incidence of severe adverse events or severe malaria in the treatment arm.
3. To measure the cost-effectiveness and acceptability of fMDA by calculating the cost per malaria case averted for intervention and control arms.

ELIGIBILITY:
Inclusion Criteria:

1. Cluster eligibility

   * Within 8 hours transport of Iquitos
   * Incidence <250/1000 and >2 cases year prior to trial
   * Population size (<650)
2. Chloroquine (CQ) eligibility

   * Resides in neighboring household but within 200 m of Pv index case in the past 2 years
   * Age ≥6 months old
   * Present for intervention
   * Adult ≥18 years old that provides informed consent
   * A child ≥8 years and <18 years old that provides informed assent and has informed consent from their parents
   * A child ≥6 months old and <8 years old that has informed consent from their parents
3. Tafenoquine (TQ) eligibility

   * Eligible to receive CQ
   * Age ≥16 years old
   * Adult ≥18 years old that provides informed consent
   * A child ≥16 years and <18 years old that provides informed assent and has informed consent from their parents
4. Primaquine eligibility

   * Eligible to receive CQ and ineligible to receive TQ
   * Age ≥6 months old
   * Adult ≥18 years old that provides informed consent
   * A child ≥8 years and <18 years old that provides informed assent and has informed consent from their parents
   * A child ≥6 months old and <8 years old that has informed consent from their parents
5. Baseline evaluation and informed consent

   -Villagers will be eligible to participate in surveys if they slept in a household in cluster randomized to control or focal mass drug administration (fMDA) for at least one night in the past four weeks
6. Eligibility for fMDA

   * High-risk villagers are defined as individuals residing in households that are within 200 meters of a Plasmodium vivax index case households from the prior 2 years (including individuals in the index case household) will be eligible to receive fMDA that cycle
   * Villagers that were eligible but missed in the 1st round in a cycle, or become eligible in the next two months, will not be eligible to receive fMDA in the 2nd round in a cycle.

Exclusion Criteria:

1. Chloroquine eligibility

   * History of retinal or visual field changes
   * Known hypersensitivity or adverse reaction to CQ
   * Currently taking CQ or have taken CQ in the past four weeks
   * Ineligible for TQ or PQ (see criteria below)
   * Hemoglobin <9 g/dL
2. Tafenoquine eligibility

   * G6PD deficiency or intermediate status (defined as activity ≤6.0 UI/gHb per SD biosensor)
   * G6PD status unknown or refusal of G6PD status test
   * Acute or severe malaria
   * Pregnancy (known or identified by pregnancy test)
   * Refusal of pregnancy test if new amenorrhea in the past 4 weeks
   * Woman breastfeeding a child that is G6PD deficient or with unknown G6PD status
   * Known hypersensitivity or adverse reaction to TQ or PQ
   * Have taken mefloquine (i.e. artesunate- mefloquine), TQ or PQ, or other antimalarial in the past four weeks
   * Hemoglobin < 9 g/dL
3. Primaquine eligibility

   * G6PD deficiency (defined as activity ≤4.0 UI/gHb per SD biosensor)
   * G6PD status unknown or refusal of G6PD status test
   * Acute or severe malaria
   * Pregnancy (known or identified by pregnancy test)
   * Refusal of pregnancy test if new amenorrhea in the past 4 weeks
   * Breastfeeding child with documented or unknown G6PD deficiency status
   * Known hypersensitivity or adverse reaction to TQ or PQ
   * Have taken mefloquine (i.e. artesunate- mefloquine), TQ or PQ, or other antimalarial in the past four weeks
   * Hemoglobin < 9 g/dL

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7530 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative Incidence of Plasmodium vivax infections | From enrollment through study completion, over 36-month follow-up study period
  Number of microscopy-confirmed, Plasmodium vivax malaria cases in residents reported from health facilities per population over the 36-month follow-up study period

SECONDARY OUTCOMES:
Prevalence of Plasmodium vivax infection | At endline survey in trial year 4, 3 years after enrollment in study in trial year 1
  Proportion of individuals with polymerase chain reaction (PCR)-confirmed infection in an endline survey
Plasmodium vivax seroprevalence | At endline survey in trial year 4, 3 years after enrollment in study in trial year 1
  Proportion of participants who are seropositive, rate at which seronegative individuals became seropositive estimated from age-specific seroprevalence from endline survey, adjusted by modeling longitudinal individual serological status and/or antibody titers
Genetic diversity of Plasmodium vivax | From enrollment through study completion, over 4 trial years
  Diversity of locally acquired infections as defined by sequencing results
Tolerability of study drugs | Over drug administration period, unique for each study drug (7 days for CQ/PQ regimens and 3 days for CQ/TQ regimens)
  Vomiting following administration of study drugs and non-adherence related to adverse effects
Adherence to study drugs | Unique for each patient based on drug regimen (7 days for CQ/PQ regimens and 3 days for CQ/TQ regimens)
  Number of missed doses
Refusal rates | During each fMDA round, twice per year for 3 consecutive years
  Number of refusals divided by number of individuals invited to participate
Program costs per unit fMDA round | From enrollment through study completion, over 4 years
  Total costs divided by number of fMDA rounds
Program costs per unit | From enrollment through study completion, over 4 years
  Total costs divided by number of individuals receiving intervention
Cost per incident case averted | From enrollment through study completion, over 4 years
  Difference in cost between fMDA and control divided by the difference in the effect (incidence)
Cost per disability life year (DALY) | From enrollment through study completion, over 4 years
  Difference in cost between fMDA and control divided by the difference in the effect (DALYs)
Cost per economic dollar due to malaria saved | From enrollment through study completion, over 4 years
  Difference in cost between fMDA and control divided by the difference in the effect (economic dollar due to malaria)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hsiang, MD, Principal Investigator — University of California, San Francisco; Alejandro Llanos-Cuentas, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Asociación Civil Selva Amazónica, Iquitos, Peru

IPD SHARING:
Plan to Share IPD: No
After completion of the trial, un-blinding will be performed and results will be disseminated widely at scientific meetings and in publications in peer-reviewed journals. Upon publication of the trial results, data will be made available for to other individuals in the scientific community upon request. Informed consent documents for the study will include a specific statement relating to posting and sharing of study information and that no individual identities will ever be used in these materials and forums.
  Human genomic data will consist of G6PD and CYP2D6 single nucleotide polymorphisms (SNPs). Plasmodium parasite genomic data will consist of microhaplotype SNPs. All genomic data will be shared in accordance with institutional and NIH policies. Informed consent forms will indicate that the investigators may share genetic data and no individual identities will be linked to these data. All genetic information generated will be analyzed through pipelines in Git.

REFERENCES:
- [Background] PAHO. Fourth Meeting of the Malaria Technical Advisory Group (TAG) to the Pan American Health Organization (PAHO). Washington D.C.: Pan American Health Organization, World Health Organization, Americas. https://www.paho.org/hq/index.php?option=com_docman&view=download&alias=50391-fourthmalaria-technical-advisory-group-meeting-report-may-washington-dc&category_slug=malariatechnical-advisory-group&Itemid=270&lang=en; 2019.
- [Background] Hsiang MS, Ntuku H, Roberts KW, Dufour MK, Whittemore B, Tambo M, McCreesh P, Medzihradsky OF, Prach LM, Siloka G, Siame N, Gueye CS, Schrubbe L, Wu L, Scott V, Tessema S, Greenhouse B, Erlank E, Koekemoer LL, Sturrock HJW, Mwilima A, Katokele S, Uusiku P, Bennett A, Smith JL, Kleinschmidt I, Mumbengegwi D, Gosling R. Effectiveness of reactive focal mass drug administration and reactive focal vector control to reduce malaria transmission in the low malaria-endemic setting of Namibia: a cluster-randomised controlled, open-label, two-by-two factorial design trial. Lancet. 2020 Apr 25;395(10233):1361-1373. doi: 10.1016/S0140-6736(20)30470-0. PMID 32334702
- [Background] Ntuku H, Smith-Gueye C, Scott V, Njau J, Whittemore B, Zelman B, Tambo M, Prach LM, Wu L, Schrubbe L, Kang Dufour MS, Mwilima A, Uusiku P, Sturrock H, Bennett A, Smith J, Kleinschmidt I, Mumbengegwi D, Gosling R, Hsiang M. Cost and cost effectiveness of reactive case detection (RACD), reactive focal mass drug administration (rfMDA) and reactive focal vector control (RAVC) to reduce malaria in the low endemic setting of Namibia: an analysis alongside a 2x2 factorial design cluster randomised controlled trial. BMJ Open. 2022 Jun 23;12(6):e049050. doi: 10.1136/bmjopen-2021-049050. PMID 35738650
- [Background] Hsiang MS, Hwang J, Tao AR, Liu Y, Bennett A, Shanks GD, Cao J, Kachur SP, Feachem RG, Gosling RD, Gao Q. Mass drug administration for the control and elimination of Plasmodium vivax malaria: an ecological study from Jiangsu province, China. Malar J. 2013 Nov 1;12:383. doi: 10.1186/1475-2875-12-383. PMID 24175930
- [Background] Llanos-Cuentas A, Lacerda MVG, Hien TT, Velez ID, Namaik-Larp C, Chu CS, Villegas MF, Val F, Monteiro WM, Brito MAM, Costa MRF, Chuquiyauri R, Casapia M, Nguyen CH, Aruachan S, Papwijitsil R, Nosten FH, Bancone G, Angus B, Duparc S, Craig G, Rousell VM, Jones SW, Hardaker E, Clover DD, Kendall L, Mohamed K, Koh GCKW, Wilches VM, Breton JJ, Green JA. Tafenoquine versus Primaquine to Prevent Relapse of Plasmodium vivax Malaria. N Engl J Med. 2019 Jan 17;380(3):229-241. doi: 10.1056/NEJMoa1802537. PMID 30650326
- [Background] World Health Organization (WHO). WHO Guidelines for malaria. 3 June 2022. https://reliefweb.int/report/world/who-guidelines-malaria-3-june-2022#:~:text=The%20WHO%20global%20malaria%20strategy,residual%20foci%20of%20malaria%20transmission.
- [Derived] Fine SR, Soto Calle V, Altamirano Quiroz A, Rodriquez Ferruci H, Manrique P, Wu X, Carrasco Escobar G, Benjamin-Chung J, Bennett A, Auburn S, Price RN, Greenhouse B, Baird JK, Domingo GJ, Roh ME, Rosas A, Llanos-Cuentas A, Hsiang MS. FocaL mass drug administration for Plasmodium vivax malaria elimination (FLAME): study protocol for an open-label cluster randomized controlled trial in Peru. Trials. 2025 Oct 14;26(1):408. doi: 10.1186/s13063-025-09112-1. PMID 41088393
- [Derived] Fine S, Quiroz AA, Calle VS, Manrique P, Rodriguez H, Carrasco G, Benjamin-Chung J, Bennett A, Auburn S, Price R, Greenhouse B, Baird JK, Domingo G, Roh M, Rosas A, Llanos-Cuentas A, Hsiang M. FocaL mass drug Administration for Plasmodium vivax Malaria Elimination (FLAME): study protocol for an open-label cluster randomized controlled trial in Peru. Res Sq [Preprint]. 2025 Apr 17:rs.3.rs-5594891. doi: 10.21203/rs.3.rs-5594891/v1. PMID 40321759